CLINICAL TRIAL: NCT01395745
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Blisibimod Administration in Subjects With Systemic Lupus Erythematosus
Brief Title: CHABLIS-SC1: A Study of the Efficacy and Safety of Subcutaneous Blisibimod in Subjects With Systemic Lupus Erythematosus
Acronym: CHABLIS-SC1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-SLE3331
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Lupus Erythematosus, Systemic; Autoimmune Diseases; A-623; Blisibimod
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- blisibimod weekly dose (Experimental)
  Interventions: Drug: blisibimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: blisibimod — blisibimod administered via subcutaneous injection every week for 52 weeks
  Arms: blisibimod weekly dose
Drug: Placebo — Placebo will be administered weekly via subcutaneous injection for 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of subcutaneous blisibimod administered in addition to standard therapy in subjects with active Systemic Lupus Erythematosus (SLE) disease as defined by SELENA-SLEDAI score ≥10 despite on-going stable corticosteroid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill at least 4 diagnostic criteria for SLE defined by American College of Rheumatology
* Positive antinuclear antibodies (ANA) and/or anti-double stranded DNA (anti-dsDNA)
* Active SLE disease as defined by SELENA-SLEDAI score ≥10 despite on-going stable corticosteroid therapy
* 18 years of age or older

Exclusion Criteria:

* Severe active vasculitis, active central nervous system lupus, active lupus nephritis, uncontrolled hypertension or poorly controlled diabetes
* Malignancy within past 5 years
* Known to be positive for HIV and/or positive at the screening visit for hepatitis B, or hepatitis C
* Liver disease
* Anemia, neutropenia, or thrombocytopenia
* Active infection requiring hospitalization or treatment with parenteral antibiotics within the past 60 days or history of repeated herpetic viral infections
* History of active tuberculosis or a history of tuberculosis infection
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving an SLE Responder Index at week 52 | Week 52

SECONDARY OUTCOMES:
Time to first severe SLE flare | Week 52
Proportion of subjects able to reduce oral steroid dose to ≤7.5 mg/day prednisone | Week 52
Change in the number of actively tender or swollen joints and in mucocutaneous disease activity | Week 52
Change in proteinuria from baseline | Week 52
Proportion of subjects with improved patient-reported outcomes | Week 52
Time to treatment failure | Week 52
Time to first renal flare | Week 52
Change from baseline in B cell subsets, anti dsDNA, C3, C4 | Week 52
Safety Profile (AEs, vital signs, labs, physical exams) | Week 52

CONTACTS AND LOCATIONS:
Locations (90):
- Belarus (5):
  - Investigator Site 603, Homyel
  - Investigator Site 604, Minsk
  - Investigator Site 601, Minsk
  - Investigator Site 605, Minsk
  - Investigator Site 602, Vitebsk
- Brazil (7):
  - Investigator Site 558, Curitiba
  - Investigator Site 555, Goiânia
  - Investigator Site 557, Juiz de Fora
  - Investigator Site 551, Porto Alegre
  - Investigator Site 559, Santo André
  - Investigator Site 554, São Paulo
  - Investigator Site 556, São Paulo
- Colombia (10):
  - Investigator Site 302, Antioquia
  - Investigator Site 303, Antioquia
  - Investigator Site 308, Atlántico
  - Investigator Site 310, Atlántico
  - Investigator Site 301, Bogotá
  - Investigator Site 311, Bogotá
  - Investigator Site 304, Cundinamarca
  - Investigator Site 305, Santander
  - Investigator Site 306, Santander
  - Investigator Site 312, Valle
- Georgia (3):
  - Investigator Site 001, Tbilisi
  - Investigator Site 002, Tbilisi
  - Investigator Site 003, Tbilisi
- Guatemala (4):
  - Investigator Site 901, Guatemala City
  - Investigator Site 902, Guatemala City
  - Investigator Site 903, Guatemala City
  - Investigator Site 904, Guatemala City
- Hong Kong (2):
  - Investigator Site 151, Pokfulam
  - Investigator Site 152, Tuenmen
- India (11):
  - Investigator Site 503, Ahmedabad
  - Investigator Site 508, Bangalore
  - Investigator Site 505, Hyderabad
  - Investigator Site 502, Hyderabad
  - Investigator Site 501, Kolkata
  - Investigator Site 506, Manipal
  - Investiagtor Site 513, Mumbai
  - Investigator Site 511, New Delhi
  - Investigator Site 512, New Delhi
  - Investigator Site 504, Pune
  - Investigator Site 510, Pune
- Malaysia (2):
  - Investigator Site 251, Kuala Selangor
  - Investigator Site 252, Perak
- Mexico (6):
  - Investigator Site 702, Guanajuato City
  - Investigator Site 703, Mexico City
  - Investigator Site 701, Mexico City
  - Investigator Site 704, Mexico City
  - Investigator Site 707, Toluca
  - Investigator Site 705, Yucatán
- Philippines (10):
  - Investigator Site 407, Angeles
  - Investigator Site 404, Cebu City
  - Investigator Site 406, Cebu City
  - Investigator Site 408, Cruz Manila
  - Investigator Site 405, Davao City
  - Investigator Site 402, Ermita, Manila
  - Investigator Site 410, Iloilo City
  - Investigator Site 401, Las Piñas
  - Investigator Site 403, Manila
  - Investigator Site 409, Manila
- Russia (12):
  - Investigator Site 052, Kemerovo
  - Investigator Site 053, Kemerovo
  - Investigator Site 054, Kursk
  - Investigator Site 051, Moscow
  - Investigator Site 058, Novosibirsk
  - Investigator Site 059, Omsk
  - Investigator Site 062, Orenburg
  - Investigator Site 057, Petrozavodsk
  - Investigator Site 056, Saint Petersburg
  - Investigator Site 061, Smolensk
  - Investigator Site 060, Vladimir
  - Investigator Site 055, Yekaterinburg
- Investigator Site 101, Singapore, Singapore
- South Korea (5):
  - Investigator Site 355, Daegu
  - Investigator Site 352, Daejeon
  - Investigator Site 353, Gwangju
  - Investigator Site 351, Jeollabuk-do
  - Investigator Site 354, Suwon
- Sri Lanka (3):
  - Investigator Site 801, Colombo
  - Investigator Site 804, Kandy
  - Investigator Site 802, Nugegoda
- Taiwan (5):
  - Investigator Site 452, Kaohsiung City
  - Investigator Site 455, Taichung
  - Investigator Site 454, Taichung
  - Investigator Site 453, Taipei
  - Investigator Site 451, Taipei
- Thailand (4):
  - Investigator Site 205, Bangkok Noi
  - Investigator Site 202, Khon Kaen
  - Investigator Site 204, Muang Chiang Mai
  - Investigator Site 201, Ratchathewi

REFERENCES:
- [Derived] Merrill JT, Shanahan WR, Scheinberg M, Kalunian KC, Wofsy D, Martin RS. Phase III trial results with blisibimod, a selective inhibitor of B-cell activating factor, in subjects with systemic lupus erythematosus (SLE): results from a randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2018 Jun;77(6):883-889. doi: 10.1136/annrheumdis-2018-213032. Epub 2018 Mar 21. PMID 29563108